CLINICAL TRIAL: NCT01749072
Title: A Phase Ⅱ Randomized Clinical Trial Comparing Vinorelbine-ifosfamide With Gefitinib as Third-line Treatment in Advanced EGFR Gene Mutation Negative Non-small Cell Lung Cancer Patients
Brief Title: Vinorelbine-ifosfamide Versus Gefitinib for EGFR Gene Mutation Negative Non-small Cell Lung Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-S464
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Non-small Cell Lung Cancer; Effects of Chemotherapy
Keywords: non small cell lung cancer; chemotherapy; gefitinib; vinorelbine; ifosfamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Vinorelbine; Ifosfamide; Mesna; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gefitinib (Other): Gefitinib group Gefitinib (Iressa) 250mg once per day until progression disease or intolerant side effects
  Interventions: Drug: Gefitinib group
- Vinorelbine-Ifosfamide (Other): VI group Vinorelbine 25mg/m2 d1,d8;Ifosfamide 1.25g/m2 d1-d3(Usually Ifosfamide 2g d1-d3 with Mesna 400mg 0,4,8hours after Ifosfamide administration for 3 days);every 3 weeks;at least for 2-6 cycles depending on the progression disease or the patient's physical condition
  Interventions: Drug: Vinorelbine, Ifosfamide, Mesna

INTERVENTIONS:
Drug: Gefitinib group — Gefitinib 250mg once per day until the progression disease or intolerant side effects
  Other Names: Gefitinib (Iressa)
  Arms: Gefitinib
Drug: Vinorelbine, Ifosfamide, Mesna — Vinorelbine 25mg/m2 d1,d8; Ifosfamide 1.25g/m1 d1-d3 (Usually 2g d1-d3); Mesna 400mg 0,4,8 hours after Ifosfamide administration for uroprotection d1-d3;
  Other Names: VI group
  Arms: Vinorelbine-Ifosfamide

SUMMARY:
In the National Comprehensive Cancer Network (NCCN) guideline for NSCLC, epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) is recommended as the third-line treatment for EGFR gene mutation negative NSCLC patients who failed to the first-line platinum doublet chemotherapy [i.e. paclitaxel-carboplatin (PC) or gemcitabine-cisplatin (GP)] and the second-line chemotherapy with docetaxel or pemetrexed. But as we know, if patients had no EGFR gene mutation, EGFR-TKI treatment is not effective. The overall survival is short and the objective response rate is low. As for EGFR gene wild type patients with good performance status, besides EGFR-TKI treatment, other first generation cytotoxic drugs i.e. vinorelbine or ifosfamide maybe an alternative treatment. So the purpose of this clinical trial is to compare the effectiveness and safety of vinorelbine-ifosfamide with gefitinib in advanced or metastatic EGFR gene mutation negative NSCLC patients.

DETAILED DESCRIPTION:
Ifosfamide is a first generation cytotoxic drug to treat NSCLC. Phase Ⅱ studies demonstrated that single-agent ifosfamide administrated by various schedules produces response rates of 15-29%, with media survival times of 5-7 months. Ifosfamide has also been used in various combination regimens to treat NSCLC, including platinum based and non-platinum regimens. But in refractory NSCLC patients platinum and some third generation cytotoxic drugs have been used before. So in this study, ifosfamide is combined with vinorelbine. In previous study, Masters reported the objective response rate was 40% and the median survival duration was 50 weeks, with a 1-year survival rate of 48% with vinorelbine-ifosfamide regimen [Vinorelbine 15 mg/m2 on days 1-3, and ifosfamide 2.0g/m2 on days 1-3 with granulocyte-colony stimulating factor (G-CSF) support]. The dose limiting toxicity (DLT) of this regimen is myelosuppression. In our experience, the regimen of vinorelbine 25mg/m2 d1, d8 and ifosfamide 1.25g/m2 d1-d3 with Mesna uroprotection is safe in Chinese population and the objective response rate is about 7% (data not published).

Gefitinib is the first small molecule inhibitor that has directed activity towards EGFR and has shown appreciable response rates in phase Ⅱ trials of patients with previously treated advanced NSCLC. In the posterior analysis of Iressa Dose Evaluation in Advanced Lung Cancer (IDEAL) and IRESSA Survival Evaluation in Lung Cancer (ISEL) trials, the response rate with gefitinib ranges from 2.6% to 10% in wild-type EGFR gene NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* age range:18-70 years old
* life expectancy more than 12 weeks
* histologically or cytologically confirmed inoperable NSCLC (stage ⅢB/Ⅳ)
* ineligible for curative radiotherapy
* no prior radiotherapy for the target lesions
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2;
* prior treatments include first-line platinum doublet chemotherapy i.e. PC or GP and second-line chemotherapy with docetaxel or pemetrexed;
* No EGFR gene mutation detected by Scorpions-ARMS;
* at least one bidimensionally measurable or radiographically assessable lesion;
* adequate bone marrow reserve;
* adequate hepatic and renal function;

Exclusion Criteria:

* prior treatments including any of the following drugs:gefitinib,vinorelbine and ifosfamide;
* additional malignancies;
* uncontrolled systemic disease;
* any evidence of clinically active interstitial lung disease;
* newly diagnosed central nervous system (CNS) metastasis and not treated by radiotherapy or surgery;
* pregnancy or breast feeding phase;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 52 weeks (about one year)
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks.

SECONDARY OUTCOMES:
Overall survival | Up to 100 weeks
  From date of randomization until the date of death from any cause, assessed up to 100 weeks.
objective response rate | up to 9 weeks
  The objective response rate includes the complete remission and partial remission rate.
the score of functional assessment of cancer treatment-lung (FACT-L) | Up to 100 weeks
  FACL-L is assessed at different time points.(Date of randomization, 1 week after chemotherapy/EGFR-TKI, every cycle of chemotherapy/EGFR-TKI, every month of EGFR-TKI treatment/observation, up to 100 weeks)
Number of participants with adverse events | Up to six months
  The adverse events are assessed by National Cancer Institute-Common Toxicity Criteria (Version 3.0) (NCI-CTC).

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Department of Respiratory Medicine, Peking Unoin Medical College Hospital
Locations (1):
- Department of Respiratory Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Thatcher N, Anderson H, Smith DB, Steward WP, Webb K, Hilton A, Rahman A. Ifosfamide by bolus as treatment for advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 1986;18 Suppl 2:S30-3. doi: 10.1007/BF00647448. PMID 3028661
- [Result] Holoye PY, Glisson BS, Lee JS, Dhingra HM, Murphy WK, Umsawasdi T, Levy JK, Jeffries D, Raber MN, Hong WK. Ifosfamide with mesna uroprotection in the management of lung cancer. Am J Clin Oncol. 1990 Apr;13(2):148-55. doi: 10.1097/00000421-199004000-00012. PMID 2156418
- [Result] Masters GA, Hoffman PC, Hsieh A, Drinkard LC, Mick R, Samuels BL, Guaspari A, Golomb HM, Vokes EE. Phase I study of vinorelbine and ifosfamide in advanced non-small-cell lung cancer. J Clin Oncol. 1997 Mar;15(3):884-92. doi: 10.1200/JCO.1997.15.3.884. PMID 9060524
- [Result] Bell DW, Lynch TJ, Haserlat SM, Harris PL, Okimoto RA, Brannigan BW, Sgroi DC, Muir B, Riemenschneider MJ, Iacona RB, Krebs AD, Johnson DH, Giaccone G, Herbst RS, Manegold C, Fukuoka M, Kris MG, Baselga J, Ochs JS, Haber DA. Epidermal growth factor receptor mutations and gene amplification in non-small-cell lung cancer: molecular analysis of the IDEAL/INTACT gefitinib trials. J Clin Oncol. 2005 Nov 1;23(31):8081-92. doi: 10.1200/JCO.2005.02.7078. Epub 2005 Oct 3. PMID 16204011
- [Result] Hirsch FR, Varella-Garcia M, Bunn PA Jr, Franklin WA, Dziadziuszko R, Thatcher N, Chang A, Parikh P, Pereira JR, Ciuleanu T, von Pawel J, Watkins C, Flannery A, Ellison G, Donald E, Knight L, Parums D, Botwood N, Holloway B. Molecular predictors of outcome with gefitinib in a phase III placebo-controlled study in advanced non-small-cell lung cancer. J Clin Oncol. 2006 Nov 1;24(31):5034-42. doi: 10.1200/JCO.2006.06.3958. PMID 17075123